CLINICAL TRIAL: NCT06487702
Title: Fruquintinib Combined With AK104 and Tegafur Gimeracial and Oteracil as Second-ine or After Line Treatment in Advanced or Metastatic ESCC
Brief Title: A Phase lb/lI Clinical Study in Advanced or Metastatic Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rui-hua Xu, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Rui-hua Xu, MD, PhD, Chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-E102
Record Dates: First submitted 2024-06-13; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — potassium oxonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental:fruquintinib+Candonilimab + Tegafur，Gimeracil and Oteracil Potassium (Experimental): Fruquintinib administration for 2 weeks followed by 1-week break
  Candonilimab：10 mg/kg，D1，Q3W；
  Tegafur，Gimeracil and Oteracil Potassium：30mg BID for body surface area < 1.25 m2; 40mg BID for body surface area of 1.25-1.5 m2; and 50mg BID for body surface area >1.5 m2; D1-14, q3w
  Interventions: Drug: fruquintinib++Candonilimab+ Tegafur，Gimeracil and Oteracil Potassium

INTERVENTIONS:
Drug: fruquintinib++Candonilimab+ Tegafur，Gimeracil and Oteracil Potassium — Fruquintinib administration for 2 weeks followed by 1-week break
  Candonilimab：10 mg/kg，D1，Q3W；
  Tegafur，Gimeracil and Oteracil Potassium：30mg BID for body surface area < 1.25 m2; 40mg BID for body surface area of 1.25-1.5 m2; and 50mg BID for body surface area >1.5 m2; D1-14, q3w

SUMMARY:
This is a prospective, single-arm, open-label，multi-center, phase Ib/II study, aiming to evaluate the efficacy and safety of Fruquintinib combined With Cadonilimab (AK104) and Tegafur，Gimeracil and Oteracil Potassium in patients with locally advanced or metastatic esophageal squamous cell carcinoma after the failure of first-line treatments.

DETAILED DESCRIPTION:
Esophageal cancer is a malignant tumor with high incidence and death rate in the world, especially in china, and Esophageal squamous cell carcinoma (ESCC) is the main pathological type of esophageal carcinoma in China. Among patients with advanced or metastatic esophageal squamous cell carcinoma, the addition of immunotherapy to chemotherapy, compared with chemotherapy, significantly improved overall survival and progression-free survival in first-line treatments. Treatment of recurrent or metastatic esophageal squamous cell carcinoma is usually poor. New treatments were needed.Fruquintinib is an orally antiangiogenic agents, which target VEGFR1/2/3. Candonilimab (AK104) is a PD-1/CTLA-4 Bispecific Antibody. A combination of Fruquintinib and Candonilimab (AK104) and s-1 for advanced or metastatic esophageal squamous cell carcinoma could be a novel therapy. Therefore, investigators initialize this phase Ib/II study to explore the efficacy and safety of fruquintinib in combination with Candonilimab (AK104) and S-1 treatment in ESCC patients with after failure in 1st-line treatment.

In dose escalation period, 3-12 patients with Esophageal squamous cell carcinoma will be enrolled. Patients meeting enrollment eligibility will receive 21-day cycles of fruquintinib 2-3 mg qd，D1-14,Q3W； combined with Candonilimab 10 mg/kg，D1，Q3W and S-1 (30mg BID for body surface area <1.25 m2;40mg BID for body surface area ≥1.25 - <1.5 m2;50mg BID for body surface area ≥1.5m2 ；D1-14,Q3W)

Safety information will be collected till disease progression or intolerable toxicity to determine MTD and/or RPTD of fruquintinib combined with Candonilimab and S-1 in patients with Esophageal squamous cell carcinoma .

This period will include the following 2 dose groups from low to high:

A: Fruquintinib 2 mg qd for 2 weeks followed by 1-week break + Candonilimab 10 mg/kg，intravenous infusion，D1, every 3 weeks+ S-1 ,Calculate dosage based on body surface ,30mg for BSA <1.25 m2;40 mg for BSA ≥1.25 - <1.5 m2; 50mg for BSA ≥1.5m2;BID，D1-14，Q3W

B: Fruquintinib 3 mg qd for 2 weeks followed by 1-week break + Candonilimab 10 mg/kg，intravenous infusion，D1, every 3 weeks+ S-1 ,Calculate dosage based on body surface ,30mg for BSA <1.25 m2;40 mg for BSA ≥1.25 - <1.5 m2; 50mg for BSA ≥1.5m2;BID，D1-14，Q3W

This study will use traditional 3+3 trial design (3 subjects will be enrolled in each dose group first).

If 1 case of DLT is observed, additional 3 subjects will be enrolled in the same dose group,when no new DLTs occurred, the trial was continued to the next dose level to further evaluate toxicity ,to observe DLT and evaluate MTD.

If there are 2 or more cases of DLT in one dose group, the group lower than this dose group by one level is MTD dose group. If 2 dose group levels MTD was not reached, then the B group dose was RP2D.(DLT was predefined by the investigator in the protocol)

Subjects in the original dose group will continue to receive the next cycle of treatment at the original dose till disease progression or treatment withdrawal due to any of the following reasons: 1) death, 2) intolerable toxicity, 3) pregnancy, 4) the investigator considers the study should be terminated for the subject's best interests, 5) the subject or legal representative requests withdrawal, 6) loss to follow-up, 7) the subject has poor compliance and cannot comply with the study protocol.

In phase II period,patients meeting enrollment eligibility will receive Fruquintinib PR2D in combination with Candonilimab 10 mg/kg，intravenous infusion，D1, every 3 weeks and S-1 ,Calculate dosage based on body surface ,30mg for BSA <1.25 m2;40 mg for BSA ≥1.25 - <1.5 m2; 50mg for BSA ≥1.5m2;BID，D1-14，Q3W, till disease progression or treatment withdrawal due to any of the following reasons: 1) death, 2) intolerable toxicity, 3) pregnancy, 4) the investigator considers the study should be terminated for the subject's best interests, 5) the subject or legal representative requests withdrawal, 6) loss to follow-up, 7) the subject has poor compliance and cannot comply with the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. age:18-75 years old, Male or female patients
2. Histologically or cytologically confirmed esophageal squamous cell carcinoma (including the gastroesophageal junction), (Adenosquamous carcinoma with squamous cell carcinoma components-based is allowed to be included)
3. Irretrievably resected, local advanced, relapsed or metastatic esophageal squamous cell carcinoma
4. Previously received platinum-based systemic anti-tumor first-line therapy; Or received Neoadjuvant, adjuvant therapy, or radical chemoradiotherapy for ESCC, but disease recurrence or progression within 6 months after completion of treatment; no restrictions on prior immunotherapy treatment choice.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 to 1
6. At least one measurable lesion (RECIST1.1)
7. Life expectancy of more than 3 months;
8. Women of childbearing age were required to have had a negative pregnancy test (serum or urine) within 14 days before enrollment and to voluntarily use an appropriate method of contraception during the observation period and for 8 weeks after the last dose of the study drug.For men, either surgical sterilization or consent to use an appropriate method of contraception during the observation period and for 8 weeks after the last dose of the study drug was given
9. Have fully understood and voluntarily sign the ICF for this study;
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure;
11. Adequate hepatic, renal, heart, and hematologic functions

Exclusion Criteria:

1. Have had other malignancies within the past 5 years, except for curatively treated radical skin basal cell or squamous cell carcinoma, Or cervical carcinoma in situ;
2. Have received major surgical procedures (such as craniotomy, thoracotomy, or laparotomy) within 4 weeks before enrollment or are excepted to uddergo major surgery during the study treatment; received laparoscopic exploration within 2 weeks before enrollment; received central venous catheterization within 7 days prior to enrollment
3. Have received chemotherapy, targeted therapy, traditional Chinese herbal medicine with anti-tumor indications or immunomodulatory drugs (including thymosin, interferon, interleukins, etc.) within the first 4 weeks prior to enrollment, or are still within 5 half-lives of such medications
4. Have symptomatic central nervous system metastases (with stable brain metastases confirmed by imageology for more than 3 months were eligible)
5. Severe infection ((≥CTCAE grade 2 infection) occurred within 4 weeks before the first dose of study drug, such as severe pneumonia requiring hospitalization, bacteremia, and infectious complications;Baseline chest imaging suggested active pulmonary inflammation with clinically relevant symptoms or signs;the presence of signs and symptoms of infection within 2 weeks before the first dose of the study drug ,or the need for treatment with oral or intravenous antibiotics was excluded if prophylactic antibiotics were used;
6. Previous and current presence of interstitial pneumonia, pneumoconiosis, drug-related pneumonia, and severely impaired pulmonary function may interfere with the detection and management of suspected drug-related pulmonary toxicity in subjects;Subjects with radiation pneumonitis within 6 months
7. Had active pulmonary tuberculosis by medical history or CT examination, or who had a history of active pulmonary tuberculosis within 1 year before enrollment ,or who had a history of active pulmonary tuberculosis more than 1 year before enrollment but had not received regular treatment
8. Congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA above the detection limit of the assay) or co-infection with hepatitis B and C;
9. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
10. With thrombotic diseases or receiving anticoagulant drugs;
11. Patients at risk of gastrointestinal hemorrhage or obstruction;
12. Unable to swallow the experimental drug;
13. Patients who have previously experienced immune-related myocarditis, pneumonitis, colitis, hepatitis, nephritis, etc.were judged to be at greater risk for immunotherapy retreatment by the investigator;
14. Patients with complications who require long-term use of immunosuppressive drugs or those who need systemic or local administration of corticosteroids with immunosuppressive effects
15. Patients considered unsuitable for inclusion in this study by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2026-06-10 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
MTD and/or PR2D | During the first 3 weeks
  To determine the Maximum Tolerated Dose ( MTD) and/or PR2D of fruquintinib combined with Cadonilimab and Tegafur,Gimeracil and Oteracil Porassium in patients with Esophageal squamous cell carcinoma (Phase Ib)
16-Week Progression-free Survival (PFS) Rate (Phase II) | 16 week
  16-Week Progression-free survival (PFS) rate is defined as the percentage of patients who are progression-free (stable disease, partial response, or complete response as defined by RECIST v1.1 criteria) at 16 weeks post registration

SECONDARY OUTCOMES:
Overall Response Rate (ORR) (Phase Ib） | Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
  from treatment up to progressive disease or EOT due to any cause up to 1 year
Disease control rate (DCR) (Phase Ib） | from treatment up to progressive disease or EOT due to any cause up to 1 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Overall survival (OS) （Phase Ib) | up to approximately 1 year
  Baseline to measured date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No